CLINICAL TRIAL: NCT05734430
Title: Genetics of Appendix Cancer: The GAP Study
Brief Title: Genetics of Appendix Cancer Study
Acronym: GAP
Status: Recruiting | Type: Observational
Sponsor: Andreana Holowatyj, PhD, MSCI (Other)
Responsible Party: Sponsor-Investigator, Andreana Holowatyj, PhD, MSCI, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Other Study IDs: VICC GI 2280
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Appendix Cancer; Appendiceal Cancer; Appendiceal Neoplasms; Appendiceal Mucinous Neoplasm; Appendiceal Adenocarcinoma; Appendiceal Carcinoid Tumor; Appendiceal Neoplasm Malignant Secondary; Appendix Adenocarcinoma; Appendix Mucinous Neoplasm; Appendix Tumor; Appendix Cancer Metastatic; Appendix NET; Low-Grade Appendix Mucinous Neoplasm; High Grade Appendix Mucinous Neoplasm; High Grade Appendix Mucinous Adenocarcinoma
Keywords: Genetics
MeSH Terms: conditions — Appendiceal Neoplasms; Adenocarcinoma, Mucinous | interventions — DNA Fingerprinting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GAP Social: Individuals ages 18+ years with an appendix cancer diagnosis in the United States.
  Interventions: Genetic: Genetic profiling; Other: Retrospective tissue procurement
- GAP Vanderbilt: Individuals ages 18+ years with an appendix cancer diagnosis seen at Vanderbilt.
  Interventions: Genetic: Genetic profiling; Other: Retrospective tissue procurement
- GAP Parent: Biological parents of active GAP (Social and Vanderbilt) Study participants.
  Interventions: Genetic: Genetic profiling

INTERVENTIONS:
Genetic: Genetic profiling — Whole exome sequencing
Other: Retrospective tissue procurement — Collection of archived fixed-formalin, paraffin-embedded (FFPE) primary appendix tumor tissues that were previously removed
  Groups: GAP Social; GAP Vanderbilt

SUMMARY:
The GAP Study is a prospective cohort study designed to comprehensively investigate genetic variations that may contribute to cancer development among individuals diagnosed with appendix/appendiceal cancer who are ages 18+ years.

DETAILED DESCRIPTION:
The Genetics of Appendix Cancer (GAP) Study aims to analyze hereditary factors, tumor characteristics and clinical features/outcomes among adults diagnosed with appendix cancer and their biological parents. Patients are recruited at any time after a diagnosis of appendix cancer and followed for up to 6 years after study enrollment. This cohort is enriched by robust biospecimens and data collections.

ELIGIBILITY:
Inclusion Criteria:

GAP Social

* Known diagnosis of appendix cancer in the United States
* Mentally and physically able to consent and participate in the study

GAP Vanderbilt

* Known diagnosis of appendix cancer
* Diagnosed by and/or consulting with a physician/clinical provider participating in the GAP Study
* Mentally and physically able to consent and participate in the study

GAP Parent

* Biological parents (mother and/or father) of individuals actively participating in the GAP Study
* Residing in the United States
* Mentally and physically able to consent and participate in the study

Exclusion Criteria:

* Women pregnant at the time of consent
* Prisoners
* Unable to provide informed consent
* Unable to read, write, or complete questionnaires in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals age 18+ years diagnosed with appendix cancer, and biological parents of study participants.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence and spectrum of pathogenic and likely pathogenic germline variants in appendix cancer patients and their biological parents | Within 6 years of study enrollment

SECONDARY OUTCOMES:
Association of germline genetic variants with clinical, pathologic and molecular features of appendix tumors | Within 6 years of study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Andreana N Holowatyj, PhD, MSCI, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Holowatyj AN, Washington MK, Tavtigian SV, Eng C, Horton C. Inherited Cancer Susceptibility Gene Sequence Variations Among Patients With Appendix Cancer. JAMA Oncol. 2022 Nov 11;9(1):95-101. doi: 10.1001/jamaoncol.2022.5425. Online ahead of print. PMID 36368039
- [Background] Holowatyj AN, Overman MJ, Votanopoulos KI, Lowy AM, Wagner P, Washington MK, Eng C, Foo WC, Goldberg RM, Hosseini M, Idrees K, Johnson DB, Shergill A, Ward E, Zachos NC, Shelton D; Appendix Cancer Pseudomyxoma Peritonei (ACPMP) Research Foundation. Defining a 'cells to society' research framework for appendiceal tumours. Nat Rev Cancer. 2025 Apr;25(4):293-315. doi: 10.1038/s41568-024-00788-2. Epub 2025 Feb 20. PMID 39979656
- [Background] Janczewski LM, Browner AE, Cotler JH, Nelson H, Kakar S, Carr NJ, Hanna NN, Holowatyj AN, Goldberg RM, Washington MK, Asare EA, Overman MJ; American Joint Committee on Cancer Expert Panel on Cancers for the Lower Gastrointestinal Appendix Disease Site. Survival outcomes used to validate version 9 of the American Joint Committee on Cancer staging system for appendiceal cancer. CA Cancer J Clin. 2023 Nov-Dec;73(6):590-596. doi: 10.3322/caac.21806. Epub 2023 Jun 26. PMID 37358310
- See also: GAP Study Website — https://www.gapcancerstudy.org